CLINICAL TRIAL: NCT01688063
Title: A Pilot Study of Skin Elasticity Measurements of the Face and Surgical Scars Stratified by Age and Skin Type
Brief Title: Skin Elasticity Measurements of the Face and Surgical Scars Stratified by Age and Skin Type
Status: Active, not recruiting | Type: Observational
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Murad Alam, Professor in Dermatology, Otolaryngology - Head and Neck Surgery, and Surgery-Organ Transplantation, Northwestern University
Other Study IDs: STU49554
Record Dates: First submitted 2011-08-15; First posted 2012-09-19 (Estimated); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Skin Scarring; Skin Elasticity
Keywords: Skin Elasticity; Scar Elasticity; Cutometer; Dermal Torque Meter
MeSH Terms: conditions — Cicatrix

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Part A: 3 Arms: Subjects will be recruited and enrolled to fill one of three Arms. The first Arm will include 25 subjects who are scheduled to receive resurfacing or tightening procedures AS STANDARD OF CARE (CO2 resurfacing or tightening procedure (1 treatment), radiofrequency (2 tx), Fraxel ( 2 tx), or PDL. These subjects will have baseline elasticity measurements recorded on their face and right forearm before their procedures, and follow up measurements will be repeated 3 months following their last treatment. The second Arm will include 25 subjects who are not scheduled to receive any cosmetic procedures but who agree to return for repeated measurements 3 months following the first. Baseline elasticity measurements will be recorded from subjects' face and right forearm and subjects will return in 3 months for follow-up measurements. The third Arm will include the remaining 50 subjects; these subjects will have the elasticity measurements performed only once on their face and forearm.
- Part B: The study population in the second cohort will consist of 250 subjects who have a surgical scar >2 cm in length. Subjects enrolled will have three elasticity measurements performed in one study visit. Elasticity will be measured directly in the center of the scar, 3cm perpendicular to the center of the scar, and 3cm in line from one end of the scar (Appendix 2).

SUMMARY:
The primary objective of Part A is to compare the change in elasticity measurements at baseline and at 3 months between subjects who have had a resurfacing or tightening procedure and those who have not. The secondary objective for Part A is to develop baseline elasticity scores for ages 18-35, 36-50, and 51-65 and for Fitzpatrick skin types I-II, III-IV, and V-VI. The primary objective of Part B is to compare the age of the scar and surrounding tissue with the elasticity measurements.

ELIGIBILITY:
Inclusion Criteria:

Part A:

* Subject is 18-65 years of age
* Subject scheduled to have resurfacing or tightening procedure done as Standard of Care (Arm 1, 25 subjects).
* The subject has the willingness and the ability to understand and provide informed consent for the use of their tissue and communicate with the investigator

Part B:

* Subject is 18 and over
* Subject has a linear surgical scar that is > 2cm.
* The subject has the willingness and the ability to understand and provide informed consent for the use of their tissue and communicate with the investigator

Exclusion Criteria:

Part A, Group 1:

-Subject is planning on having a cosmetic procedure done to their face during the 3 months they are participating in the study (Arm 2, 25 subjects).

Parts A and B:

* Under 18 years of age
* Pregnancy or Lactation
* Subjects who are unable to understand the protocol or to give informed consent
* Subjects with mental illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Up to 350 subjects who meet the inclusion/exclusion criteria for either study Part A, Part B or both will be consented and enrolled with the goal of having 100 subjects complete Part A and 250 subjects complete Part B. Subjects will be recruited from the Dermatology Clinic at Northwestern University and other Northwestern University clinics.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2011-07; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Skin elasticity measurement of participant's scars | up to 3 months
  Difference in skin elasticity measurements will be compared between subjects of varying ages at different anatomical sites: scarred sites, forehead, cheeks, mandible, and inner arm.

CONTACTS AND LOCATIONS:
Overall Officials: Murad Alam, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Feinberg School of Medicine, Department of Dermatology, Chicago, Illinois, United States